CLINICAL TRIAL: NCT04968847
Title: LOCAL: Prospective Multi-Center LOCALized Directional Insemination Trial for Artificial Insemination
Brief Title: FemaSeed LOCAL Artificial Insemination Trial
Acronym: LOCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Femasys Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-200-001
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Infertility; Male Factor
Keywords: Infertility; IUI; Intrauterine Insemination; Unexplained; Male; Sperm
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Device: FemaSeed Localized Directional Insemination (Experimental): FemaSeed (Intratubal Insemination - K231730)
  Interventions: Device: FemaSeed Localized Directional Insemination

INTERVENTIONS:
Device: FemaSeed Localized Directional Insemination — Subjects undergoing FemaSeed Artificial Insemination

SUMMARY:
Brief Summary: The objectives of the trial are to evaluate the safety and effectiveness of the FemaSeed Localized Directional Insemination for artificial insemination, now known as the FemaSeed Intratubal Insemination since FDA Cleared under K231730 in September 2023.

DETAILED DESCRIPTION:
314 subjects enrolled (signed inform consent) inclusive of 188 subjects in protocol versions 1-4 and 126 subjects in protocol version 5 (including re-consented subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Female, 19-40 years of age, with no tubal, uterine or ovarian infertility factor (including patent fallopian tubes with no evidence of hydrosalpinx)

Exclusion Criteria:

1. Greater than three prior intrauterine insemination (IUI) cycles
2. Current or recent (within the last 3 months) pelvic infection (cervix, endometrium, or fallopian tubes)
3. Prior history of ectopic pregnancy or tubal surgery

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 314 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Confirmed pregnancy rate at approximately 3 weeks following FemaSeed procedure. | 3 weeks
  Confirmed pregnancy rate per cycle: defined as the proportion of cycles with one intrauterine insemination with FemaSeed that result in pregnancy.
Primary Safety: Occurrence of ectopic pregnancy per cycle | 7 weeks
  Occurrence of ectopic pregnancy per cycle: defined as the proportion of cycles with one intrauterine insemination with FemaSeed that result in a definitively confirmed ectopic pregnancy (based on current accepted clinical standards)
Primary Safety: Occurrence of uterine perforation per cycle | At time of procedure
  Occurrence of uterine perforation per cycle: defined as the proportion of cycles with one intrauterine insemination with FemaSeed that result in uterine perforation.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Elite IVF, PLLC, Mobile, Alabama
  - Reproductive Associates of Delaware (RAD Fertility), Newark, Delaware
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Saginaw Valley Medical Research Group, Saginaw, Michigan
  - The Fertility Center of Las Vegas, Las Vegas, Nevada
  - Red Rock Fertility Center, Las Vegas, Nevada
  - Reach Fertility, Charlotte, North Carolina
  - Carolina Conceptions, Raleigh, North Carolina
  - Institute for Reproductive Health, Cincinnati, Ohio
  - University of Cincinnati Physicians, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Main Line Fertility, Bryn Mawr, Pennsylvania
  - University of Pennsylvania (Pennsylvania Fertility Care), Philadelphia, Pennsylvania
  - LinQ Research, Sugar Land, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Utah Center for Reproductive Medicine, Salt Lake City, Utah
  - University of Wisconsin, Generations Fertility Care, Middleton, Wisconsin

IPD SHARING:
Plan to Share IPD: No